CLINICAL TRIAL: NCT02499783
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Adalimumab for the Induction and Maintenance of Clinical Remission in Chinese Patients With Moderately to Severely Active Crohn's Disease and Elevated High-Sensitivity C-reactive Protein
Brief Title: Study to Evaluate the Safety and Efficacy of Adalimumab in Chinese Subjects With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-233
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-05

CONDITIONS: Crohn's Disease
Keywords: China; Tumor necrosis factor (TNF)-alpha; Biologic
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Induction Regimen (Experimental): Double-blind period (Weeks 0-8): Placebo at Weeks 0 and 2, followed by adalimumab 160 mg at Week 4, 80 mg at Week 6.
  Open label period: adalimumab 40 mg every other week (eow) from Week 8 through last dose at Week 24.
  Interventions: Biological: adalimumab; Other: placebo
- Adalimumab Induction Regimen (Experimental): Double-blind period (Weeks 0-8): adalimumab 160 mg at Weeks 0 and 80 mg at Week 2, followed by adalimumab 40 mg at Week 4 and Week 6.
  Open label period: adalimumab 40 mg eow from Week 8 through last dose at Week 24.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — subcutaneous injections of adalimumab
  Other Names: Humira
Other: placebo — subcutaneous injections of placebo
  Arms: Placebo Induction Regimen

SUMMARY:
This study will evaluate the efficacy and safety of adalimumab induction and maintenance treatment in subjects with moderately to severely active Crohn's disease in China.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of Chinese descent with full Chinese parentage.
* Diagnosis of Crohn's disease (CD) for at least 3 months prior to Week 0.
* Crohn's Disease Activity Index (CDAI) greater than or equal to 220 and less than or equal to 450 despite treatment with oral corticosteroids and/or immunosuppressants.
* Subject has a negative Tuberculosis (TB) Screening Assessment.
* Subject has elevated high sensitivity C-reactive protein (hs-CRP) during the Screening Period.

Exclusion Criteria:

* Subject with ulcerative colitis or indeterminate colitis.
* Subject who has had a surgical bowel resection within the past 6 months or who is planning any resection at any time point in the future.
* Subject with an ostomy or ileoanal pouch.
* Subject who has short bowel syndrome.
* Subject with symptomatic known obstructive strictures.
* Subject with an internal or external fistula (with the exception of an anal fistula without abscess).
* Active, or chronic or recurring infections, or active tuberculosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen B, Gao X, Zhong J, Ren J, Zhu X, Liu Z, Wu K, Kalabic J, Yu Z, Huang B, Kwatra N, Doan T, Robinson AM, Chen MH. Efficacy and safety of adalimumab in Chinese patients with moderately to severely active Crohn's disease: results from a randomized trial. Therap Adv Gastroenterol. 2020 Jul 16;13:1756284820938960. doi: 10.1177/1756284820938960. eCollection 2020. PMID 32733600

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-Blind (DB) Period: Adalimumab 160/80/40 mg: Double-blind adalimumab 160 mg at Week 0; 80 mg at Week 2; 40 mg at Weeks 4 and 6.
- DB Period: Placebo Followed by Adalimumab 160/80 mg: Double-blind placebo at Weeks 0 and 2, adalimumab 160 mg at Week 4, 80 mg at Week 6.
- Open-Label (OL) Period: Adalimumab 40 mg: Open-label adalimumab 40 mg every other week (eow) from Week 8 through last dose at Week 24.
Period: DB Period/Placebo-Controlled: Weeks 0-4
Arm/Group | Double-Blind (DB) Period: Adalimumab 160/80/40 mg | DB Period: Placebo Followed by Adalimumab 160/80 mg | Open-Label (OL) Period: Adalimumab 40 mg
Started | 102 | 103 | 0
Completed | 98 | 98 | 0
Not Completed | 4 | 5 | 0
Not completed — Adverse Event | 2 | 4 | 0
Not completed — Withdrew Consent | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0
Period: DB Period: Weeks 0-8
Arm/Group | Double-Blind (DB) Period: Adalimumab 160/80/40 mg | DB Period: Placebo Followed by Adalimumab 160/80 mg | Open-Label (OL) Period: Adalimumab 40 mg
Started | 102 | 103 | 0
Completed | 92 | 96 | 0
Not Completed | 10 | 7 | 0
Not completed — Adverse Event | 8 | 6 | 0
Not completed — Withdrew Consent | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0
Period: Open Label Period: Weeks 8 to 26
Arm/Group | Double-Blind (DB) Period: Adalimumab 160/80/40 mg | DB Period: Placebo Followed by Adalimumab 160/80 mg | Open-Label (OL) Period: Adalimumab 40 mg
Started | 0 | 0 | 188
Completed | 0 | 0 | 159
Not Completed | 0 | 0 | 29
Not completed — Adverse Event | 0 | 0 | 16
Not completed — Withdrew Consent | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 9
Not completed — Subject Noncompliance | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Double-Blind Period: Adalimumab 160/80/40 mg: Double-blind adalimumab 160 mg at Week 0; 80 mg at Week 2; 40 mg at Weeks 4 and 6.
- Double-Blind Period: Placebo Followed by Adalimumab 160/80 mg: Double-blind placebo at Weeks 0 and 2, adalimumab 160 mg at Week 4, 80 mg at Week 6.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period: Adalimumab 160/80/40 mg | Double-Blind Period: Placebo Followed by Adalimumab 160/80 mg | Total
Number analyzed (Participants) | 102 | 103 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.24) | 32.6 (9.50) | 32.9 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 65
  Male | 67 | 73 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 102 | 103 | 205
Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — CDAI is used to quantify the symptoms of subjects with Crohn's Disease. It generally ranges from 0 up to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
  units on a scale | 272.05 (48.117) | 274.71 (49.055) | 273.38 (48.490)
High Sensitivity C-Reactive Protein (Hs-CRP) [Mean (Standard Deviation); unit: mg/L] | 23.93 (24.595) | 27.12 (31.526) | 25.53 (28.266)
Fecal Calprotectin [Mean (Standard Deviation); unit: μg/g] | 1481.8 (809.29) | 1435.4 (766.37) | 1458.4 (786.20)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) at Week 4
Description: CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 4
Population: Intention to Treat (ITT) Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Double-Blind Period, Weeks 0 to 4: Placebo: Double-blind placebo at Weeks 0 and 2
- Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg: Double-blind adalimumab 160 mg at Week 0 and 80 mg at Week 2
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 6.8 | 37.3
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Stratified by Crohn's disease severity (CDAI <= 300 and CDAI >300) at baseline and corticosteroid use at baseline; Adjusted Risk Difference = 30.4, 95% CI 2-sided [19.2 to 41.7] — Risk difference = (adalimumab 160/80 mg - placebo). Stratified by Crohn's disease severity (CDAI <= 300 and CDAI >300) at baseline and corticosteroid use at baseline

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 26 (CDAI < 150) in Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 8
Description: as for outcome 1
Time Frame: Week 26
Population: All participants who were randomized and who achieved clinical response (decrease in CDAI ≥ 70 points from Baseline) at Week 8. Non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Double-blind period: placebo at Weeks 0 and 2, adalimumab 160 mg at Week 4, 80 mg at Week 6, OR Double-blind period: adalimumab 160 mg at Week 0, 80 mg at Week 2, 40 mg at Weeks 4 and 6.
  Open label period: adalimumab 40 mg eow from Week 8 through last dose at Week 24.
Arm/Group | All Participants
Number analyzed (Participants) | 144
percentage of participants | 64.6
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.001, One Sample Exact Test; The one sample Exact test was performed by comparing it to the clinically meaningful remission rate of 30%; Risk Difference Compared to 30% = 34.6, 95% CI 2-sided [26.2 to 42.4]

3. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Plus a Reduction in Hs-CRP of at Least 50% From Baseline at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 0 | 33.3
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by be stratified by Crohn's disease severity (CDAI <= 300, > 300) at Baseline and corticosteroid use at Baseline; Adjusted Risk Difference = 33.4, 95% CI 2-sided [23.2 to 43.6] — Risk difference = (adalimumab 160/80 mg - placebo). Based on Cochran-Mantel-Haenszel test stratified by be stratified by Crohn's disease severity (CDAI <= 300, > 300) at Baseline and corticosteroid use at Baseline

4. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Plus a Reduction in Hs-CRP of At Least 50% From Baseline at Week 26 in Participants Who Achieved Clinical Response Plus at Least 30% Reduction in Hs-CRP From Baseline at Week 8
Description: Clinical response is defined as a decrease in CDAI ≥ 70 Points from Baseline
  CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 26
Population: All participants who were randomized and who achieved clinical response (decrease in CDAI ≥ 70 points from Baseline) plus at least 30% reduction in hs-CRP from Baseline at Week 8. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 120
percentage of participants | 55.0

5. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroid Use and Achieved Clinical Remission at Week 26 in Participants Who Were Taking Steroids at Baseline and Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 8
Description: as for outcome 1
Time Frame: Week 26
Population: All participants who were randomized and who were taking steroids at Baseline and who achieved clinical response (decrease in CDAI ≥ 70 points from Baseline) at Week 8. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 43
percentage of participants | 62.8

6. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroid Use and Achieved CDAI < 150 Plus a Reduction in Hs-CRP of ≥ 50% From Baseline (BL) at Week 26 in Participants Taking Steroids at BL and Who Achieved CDAI Decrease and Hs-CRP Reduction at Week 8
Description: Percentage of participants who discontinued corticosteroid use and achieved clinical remission (CDAI < 150) plus a reduction in hs-CRP of at least 50% from Baseline at Week 26 in participants who were taking steroids at Baseline and who achieved clinical response (decrease in CDAI of ≥ 70 points from Baseline) plus a reduction in hs-CRP of ≥ 30% From Baseline at Week 8.
  CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 26
Population: All participants who were randomized and who were taking steroids at Baseline and who achieved clinical response (decrease in CDAI ≥ 70 points from Baseline) plus a reduction in hs-CRP of at least 30% from Baseline at Week 8. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 33
percentage of participants | 57.6

7. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 27.2 | 67.6
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Adjusted Risk Difference = 40.4, 95% CI 2-sided [26.7 to 54.2] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) Plus a Reduction in Hs-CRP of at Least 30% From Baseline at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 11.7 | 61.8
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Adjusted Risk Difference = 50.2, 95% CI 2-sided [36.9 to 63.5] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) and Hs-CRP < 3 mg/L at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 0 | 27.5
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Adjusted Risk Difference = 27.6, 95% CI 2-sided [18.2 to 37.0] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150), Hs-CRP < 3 mg/L at Week 26 in Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 8
Description: as for outcome 1
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 144
percentage of participants | 36.8

11. Secondary Outcome: Percentage of Participants Who Achieved Inflammatory Bowel Disease Questionnaire (IBDQ) Remission (IBDQ ≥ 170 Points) at Week 4
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). Total IBDQ score is the sum of the responses to the individual IBDQ questions, and ranges from 32 to 224 with higher scores indicating a better quality of life.
Time Frame: Week 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 20.4 | 40.2
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Adjusted Risk Difference = 19.6, 95% CI 2-sided [7.1 to 32.1] — [estimate comment as in outcome 3, analysis 1]

12. Secondary Outcome: Percentage of Participants Who Achieved IBDQ Remission (IBDQ ≥ 170 Points) at Week 26 in Participants With Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 8
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). Total IBDQ score is the sum of the responses to the individual IBDQ questions, and ranges from 32 to 224 with higher scores indicating a better quality of life.
  CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 144
percentage of participants | 51.4

13. Secondary Outcome: Change From Baseline in Fecal Calprotectin Level at Week 4
Time Frame: Baseline, Week 4
Population: ITT Set: all participants who were randomized. Observed cases.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 93 | 91
μg/g | -66.3 (844.89) | -499.5 (868.62)
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p < 0.001, ANCOVA — P-value for test of difference between adalimumab and placebo for mean change from Baseline using ANCOVA with Treatment, Crohn's disease severity (CDAI <= 300, > 300) at Baseline and corticosteroid use at Baseline, and Baseline value as covariate; Least Squares Mean Difference = -385.2, 95% CI 2-sided [-598.81 to -171.50]

14. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150), Hs-CRP < 3 mg/L and Fecal Calprotectin < 250 μg/g at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants | 0 | 9.8
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Adjusted Risk Difference = 9.8, 95% CI 2-sided [3.9 to 15.8] — [estimate comment as in outcome 3, analysis 1]

15. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150), Hs-CRP < 3 mg/L and Fecal Calprotectin < 250 μg/g at Week 26 in Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 8
Description: as for outcome 1
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 144
percentage of participants | 16.0

16. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Over Double-Blind Weeks 0-4
Description: CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
  The analysis over time was performed for the DB placebo-controlled period (Week 0 to Week 4), with comparisons between active treatment and placebo groups. The analysis over time was also performed for Any Adalimumab set (the entire study on or after the first dose of adalimumab), with only summary statistics for adalimumab treatment.
Time Frame: Weeks 2, 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants
  Week 2 | 7.8 | 26.5
  Week 4 | 6.8 | 37.3
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Clinical Remission at Week 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by Crohn's disease severity (CDAI <= 300 and CDAI >300) at baseline and corticosteroid use at baseline; Adjusted Risk Difference = 18.4, 95% CI 2-sided [8.2 to 28.6] — Risk difference = (adalimumab 160/80 mg - placebo). Based on Cochran-Mantel-Haenszel test stratified by Crohn's disease severity (CDAI <= 300 and CDAI >300) at baseline and corticosteroid use at baseline
Statistical Analysis 2: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Clinical Remission at Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 30.4, 95% CI 2-sided [19.2 to 41.7] — [estimate comment as in outcome 16, analysis 1]

17. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Over Time (Any Adalimumab Set)
Description: CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
  The analysis over time was performed for the DB placebo-controlled period (Week 0 to Week 4), with comparisons between active treatment and placebo groups. The analysis over time was also performed for Any Adalimumab set (the entire study on or after the first dose of adalimumab), with only summary statistics for adalimumab treatment. (Note: the analysis window for the 'Any Adalimumab Set' is different from that used for the ITT population. For the Any Adalimumab Set, the Baseline Visit date is the date when the first dose of adalimumab was received, and was counted as Day 1 or Week 0.)
Time Frame: Baseline (Week 0 of adalimumab), Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 200
percentage of participants
  Baseline | 3.0
  Week 2 | 31.5
  Week 4 | 40.0
  Week 6 | 48.0
  Week 8 | 55.5
  Week 10 | 45.5
  Week 12 | 56.5
  Week 14 | 51.5
  Week 16 | 56.0
  Week 18 | 48.5
  Week 20 | 53.0
  Week 22 | 52.5
  Week 24: number analyzed (Participants) | 102
  Week 24 | 49.0
  Week 26: number analyzed (Participants) | 102
  Week 26 | 53.9

18. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Plus A Reduction in Hs-CRP of at Least 50% From Baseline Over Double-Blind Weeks 0-4
Description: as for outcome 16
Time Frame: Weeks 2, 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants
  Week 2 | 1.0 | 22.5
  Week 4 | 0 | 33.3
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Clinical Remission (CDAI < 150) Plus A Reduction in HS-CRP of at Least 50% From Baseline at Week 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 21.4, 95% CI 2-sided [12.6 to 30.2] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Clinical Remission (CDAI < 150) Plus A Reduction in HS-CRP of at Least 50% From Baseline at Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 33.4, 95% CI 2-sided [23.2 to 43.6] — [estimate comment as in outcome 16, analysis 1]

19. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Plus a Reduction in Hs-CRP of at Least 50% From Baseline Over Time (Any Adalimumab Set)
Description: as for outcome 17
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 200
percentage of participants
  Week 2 | 27.5
  Week 4 | 36.0
  Week 6 | 26.0
  Week 8 | 45.0
  Week 12 | 43.5
  Week 16 | 44.5
  Week 20 | 42.0
  Week 26: number analyzed (Participants) | 102
  Week 26 | 39.2

20. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) Over Double-Blind Weeks 0-4
Description: as for outcome 16
Time Frame: Weeks 2, 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants
  Week 2 | 22.3 | 44.1
  Week 4 | 27.2 | 67.6
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 2; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 21.7, 95% CI 2-sided [8.7 to 34.6] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) at Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 40.4, 95% CI 2-sided [26.7 to 54.2] — [estimate comment as in outcome 16, analysis 1]

21. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) Over Time (Any Adalimumab Set)
Description: as for outcome 17
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 200
percentage of participants
  Week 2 | 45.0
  Week 4 | 59.0
  Week 6 | 60.0
  Week 8 | 64.5
  Week 10 | 54.5
  Week 12 | 58.0
  Week 14 | 54.5
  Week 16 | 58.0
  Week 18 | 49.5
  Week 20 | 54.5
  Week 22 | 50.0
  Week 24: number analyzed (Participants) | 102
  Week 24 | 52.9
  Week 26: number analyzed (Participants) | 102
  Week 26 | 59.8

22. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) Plus a Reduction in Hs-CRP of at Least 30% From Baseline Over Double-Blind Weeks 0-4
Description: as for outcome 16
Time Frame: Weeks 2, 4
Population: ITT Set: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
percentage of participants
  Week 2 | 8.7 | 40.2
  Week 4 | 11.7 | 61.8
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Decrease in CDAI ≥ 70 Points From Baseline Plus a Reduction in Hs-CRP of at Least 30% From Baseline at Week 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 31.4, 95% CI 2-sided [19.6 to 43.2] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Decrease in CDAI ≥ 70 Points From Baseline Plus a Reduction in Hs-CRP of at Least 30% From Baseline at Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Adjusted Risk Difference = 50.2, 95% CI 2-sided [36.9 to 63.5] — [estimate comment as in outcome 16, analysis 1]

23. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (Decrease in CDAI ≥ 70 Points From Baseline) Plus a Reduction in Hs-CRP of at Least 30% From Baseline Over Time (Any Adalimumab Set)
Description: as for outcome 17
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 200
percentage of participants
  Week 2 | 41.5
  Week 4 | 55.0
  Week 6 | 35.5
  Week 8 | 55.5
  Week 12 | 49.5
  Week 16 | 51.0
  Week 20 | 45.5
  Week 26: number analyzed (Participants) | 102
  Week 26 | 52.0

24. Secondary Outcome: Change From Baseline in CDAI Over Double-Blind Weeks 0-4
Description: as for outcome 16
Time Frame: Baseline, Weeks 2, 4
Population: ITT Set: all participants who were randomized. Observed cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
units on a scale
  Week 2 | -30.97 (53.699) | -73.66 (63.267)
  Week 4: number analyzed (Participants) | 101 | 101
  Week 4 | -38.22 (60.918) | -104.56 (67.325)
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Change From Baseline in CDAI at Week 2; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; Least Squares Mean Difference = -43.34, 95% CI 2-sided [-59.39 to -27.30]
Statistical Analysis 2: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Change From Baseline in CDAI at Week 4; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; Least Squares Mean Difference = -66.63, 95% CI 2-sided [-84.20 to -49.06]

25. Secondary Outcome: Change From Baseline in CDAI Over Time (Any Adalimumab Set)
Description: as for outcome 17
Time Frame: Baseline (Week 0 of adalimumab), Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Observed cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 200
units on a scale
  Week 2 | -67.31 (67.268)
  Week 4: number analyzed (Participants) | 197
  Week 4 | -92.60 (74.666)
  Week 6: number analyzed (Participants) | 184
  Week 6 | -103.62 (79.094)
  Week 8: number analyzed (Participants) | 176
  Week 8 | -115.96 (83.900)
  Week 10: number analyzed (Participants) | 146
  Week 10 | -122.51 (82.991)
  Week 12: number analyzed (Participants) | 152
  Week 12 | -131.55 (76.754)
  Week 14: number analyzed (Participants) | 135
  Week 14 | -136.85 (76.459)
  Week 16: number analyzed (Participants) | 140
  Week 16 | -143.56 (72.597)
  Week 18: number analyzed (Participants) | 125
  Week 18 | -140.40 (77.473)
  Week 20: number analyzed (Participants) | 128
  Week 20 | -147.54 (72.352)
  Week 22: number analyzed (Participants) | 127
  Week 22 | -143.99 (77.972)
  Week 24: number analyzed (Participants) | 54
  Week 24 | -182.01 (54.588)
  Week 26: number analyzed (Participants) | 62
  Week 26 | -178.74 (54.277)

26. Secondary Outcome: Change From Baseline in Hs-CRP Level Over Double-Blind Weeks 0-4
Description: The analysis over time was performed for the DB placebo-controlled period (Week 0 to Week 4), with comparisons between active treatment and placebo groups. The analysis over time was also performed for Any Adalimumab set (the entire study on or after the first dose of adalimumab), with only summary statistics for adalimumab treatment.
Time Frame: Baseline, Weeks 2, 4
Population: ITT Set: all participants who were randomized. Observed cases.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Double-Blind Period, Weeks 0 to 4: Placebo | Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg
Number analyzed (Participants) | 103 | 102
mg/L
  Week 2 | -4.149 (22.1944) | -16.474 (25.5491)
  Week 4: number analyzed (Participants) | 100 | 100
  Week 4 | -1.131 (18.8392) | -16.670 (19.9088)
Statistical Analysis 1: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Change From Baseline in hs-CRP Level at Week 2; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; Least Squares Mean Difference = -13.921, 95% CI 2-sided [-19.183 to -8.659]
Statistical Analysis 2: Comparison: Double-Blind Period, Weeks 0 to 4: Placebo vs Double-Blind Period, Weeks 0 to 4: Adalimumab 160/80 mg; Change From Baseline in hs-CRP Level at Week 4; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; Least Squares Mean Difference = -16.844, 95% CI 2-sided [-21.206 to -12.483]

27. Secondary Outcome: Change From Baseline in Hs-CRP Level Over Time (Any Adalimumab Set)
Description: The analysis over time was performed for the DB placebo-controlled period (Week 0 to Week 4), with comparisons between active treatment and placebo groups. The analysis over time was also performed for Any Adalimumab set (the entire study on or after the first dose of adalimumab), with only summary statistics for adalimumab treatment. (Note: the analysis window for the 'Any Adalimumab Set' is different from that used for the ITT population. For the Any Adalimumab Set, the Baseline Visit date is the date when the first dose of adalimumab was received, and was counted as Day 1 or Week 0.)
Time Frame: Baseline (Week 0 of adalimumab), Weeks 2, 4, 6, 8, 12, 16 20, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Observed cases.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 200
mg/L
  Week 2 | -16.923 (23.8242)
  Week 4: number analyzed (Participants) | 196
  Week 4 | -17.064 (21.8366)
  Week 6: number analyzed (Participants) | 130
  Week 6 | -12.295 (20.9586)
  Week 8: number analyzed (Participants) | 177
  Week 8 | -14.565 (18.5093)
  Week 12: number analyzed (Participants) | 157
  Week 12 | -13.527 (19.9087)
  Week 16: number analyzed (Participants) | 142
  Week 16 | -13.504 (18.1452)
  Week 20: number analyzed (Participants) | 133
  Week 20 | -11.921 (18.4776)
  Week 26: number analyzed (Participants) | 62
  Week 26 | -12.308 (14.4531)

28. Secondary Outcome: Change From Baseline in Fecal Calprotectin Level Over Time (Any Adalimumab Set)
Description: as for outcome 26
Time Frame: Baseline (Week 0 of adalimumab), Weeks 4, 8, 26
Population: Any Adalimumab Set: all participants who received at least 1 injection of adalimumab. Observed cases.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | All Participants
Number analyzed (Participants) | 188
μg/g
  Week 4 | -425.7 (940.04)
  Week 8: number analyzed (Participants) | 93
  Week 8 | -529.6 (913.50)
  Week 26: number analyzed (Participants) | 133
  Week 26 | -475.6 (978.07)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs): from first dose of study drug through last dose (Week 24) plus 70 days.
Description: A TEAE during Week 0-4 of DB period=any event with an onset date on or after first dose of study drug and up to first dose of study drug at Week 4 or within 70 days after the last dose of study drug in Week0-4 of DB period for participants who discontinued prior to Week 4.
  A TEAE during DB or OL period of Any Adalimumab=any event with an onset date on or after first dose of adalimumab in the DB/OL periods and within 70 days after the last dose of study drug.
Groups:
- Double-Blind Placebo Weeks 0-4: Double-blind placebo at Weeks 0 and 2.
- Double-Blind Adalimumab 160/80 mg Weeks 0-4: Double-blind adalimumab 160/80 mg at Weeks 0 and 2.
- Any Adalimumab: Any adalimumab, from first dose of adalimumab to last dose at Week 24.
Arm/Group | Double-Blind Placebo Weeks 0-4 | Double-Blind Adalimumab 160/80 mg Weeks 0-4 | Any Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/102 | 0/200
Serious Adverse Events (participants affected / at risk) | 1/103 | 2/102 | 36/200
Other Adverse Events (participants affected / at risk) | 18/103 | 25/102 | 137/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Placebo Weeks 0-4 (N=103) | Double-Blind Adalimumab 160/80 mg Weeks 0-4 (N=102) | Any Adalimumab (N=200)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 2
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 2
ANAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 17
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1
ILEAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL MASS (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
RECTAL POLYP (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 1
COLONIC ABSCESS (Infections and infestations) | 0 | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 0 | 1
PERITONITIS (Infections and infestations) | 0 | 0 | 2
TOXIC SHOCK SYNDROME (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 1
PITYRIASIS ROSEA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ABORTION INDUCED (Surgical and medical procedures) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Placebo Weeks 0-4 (N=103) | Double-Blind Adalimumab 160/80 mg Weeks 0-4 (N=102) | Any Adalimumab (N=200)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 3 | 22
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 10
PYREXIA (General disorders) | 4 | 1 | 15
INFLUENZA (Infections and infestations) | 1 | 2 | 13
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 1 | 23
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 4 | 20
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 3 | 1 | 13
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 6 | 39
DIZZINESS (Nervous system disorders) | 0 | 4 | 12
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 16
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT02499783/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT02499783/SAP_001.pdf